CLINICAL TRIAL: NCT07059910
Title: Prevalence of Thyroid Disorders in Patients With Immune Thrombocytopenic Purpura and Its Impact on Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayah Ibrahim Nemr, Assiut, Assiut University
Other Study IDs: ITP and thyroid disorders
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenic Purpura; Thyroid Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thyroid Diseases | interventions — Clinical Laboratory Techniques; Steroids; Inosine Triphosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients known ITP: Patients known ITP either newly diagnosed, chronic, refractory Age 18 yrs and above Patients with thyrodiectomy will not be in our study
  Interventions: Diagnostic Test: Search for thyroid disorders; Diagnostic Test: Laboratory test; Drug: Steroid and eltrombopage

INTERVENTIONS:
Diagnostic Test: Search for thyroid disorders — TSH , FT3 , FT4
  Other Names: Laboratory test
Diagnostic Test: Laboratory test — Search for anti thyroid antibodies
Drug: Steroid and eltrombopage — See when we treat thyroid disorders, will patient respond to steroid or eltrombopage?
  Other Names: Drugs used in ITP

SUMMARY:
Prevalence of thyroid disorders in patients with immune thrombocytopenic purpura and its impact on treatment

DETAILED DESCRIPTION:
We investigate patients with ITP for screening of thyroid disorders and how to deal with it and effect of this on the ttt

ELIGIBILITY:
Inclusion Criteria:

* ITP patients will be classified as newly diagnosed, persistent and chronic based on duration less than 3 months, 3-12 months, and more than 12 months respectively.

  * refractory ITP patients.

Exclusion Criteria:

* patients with history of thyroidectomy

  * patients with history of drug induced ITP
  * patients with history of HCV, HBV and HIV infection.
  * Patients who refuse to contribute in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective cross sectional study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Assess the frequency of thyroid disorders in patients with IT | Assess the frequency of thyroid disorders in patients with IT
  Screening of thyroid disorders in patients with ITP
Evaluate the treatment of thyroid disorders in improvement in platelets count. | Evaluate the treatment of thyroid disorders in improvement in platelets count.
  Evaluate if patients have managed according to thyroid disorders, will this affect in their response to ITP management